CLINICAL TRIAL: NCT03963310
Title: Evaluation and Follow-up of Optic Neuritis Not Related to Multiple Sclerosis
Brief Title: Optical Coherence Tomography and Optic Neuritis Not Related to Multiple Sclerosis
Acronym: OCTON2
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: RDS_2019_8
Record Dates: First submitted 2019-05-20; First posted 2019-05-24 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Optic Neuritis
MeSH Terms: conditions — Optic Neuritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The visual prognosis of optic neuritis not related to multiple sclerosis is unknown, both in terms of functional recovery and evolution.

This prospective cohort study aim to assess the ophthalmological evolution of patients presenting an episode of optic neuritis (NO) not related to a multiple sclerosis or to a clinically isolated syndrome.

ELIGIBILITY:
Inclusion Criteria:

* First onset of an optic neuritis lasting for less than 1 month
* With a brain MRI that does not meet the MS criteria

Exclusion Criteria:

* Contra-indication to MRI
* Pregnant or lactating woman
* History of known ipsilateral optic neuritis
* Ophthalmologic comorbidity in the ipsilateral eye that may interfere with the interpretation of the examinations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at the Adolphe de Rothschild Foundation for the first onset of an optic neuritis not related to multiple sclerosis and clinically isolated syndrome
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Visual acuity (ETDRS scale) | 1 year
  Evolution over 1 year of the ophthalmological parameters of patients treated for an episode of optic neuritis not related to multiple sclerosis or a clinically isolated syndrome
Thickness of the layers of the retina with Optical Coherent Tomography(OCT), | 1 year
Standard Humphrey Visual Field Test | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Romain DESCHAMPS, MD, Principal Investigator — Fondation A. de Rothschild
Locations (1):
- Fondation A. de Rothschild, Paris, France